CLINICAL TRIAL: NCT01155336
Title: The Effects of Lovaza® on Platelet Function and Cardiac Electrophysiology in Acute Myocardial Infarction
Brief Title: The Effects of Lovaza® in Acute Myocardial Infarction
Acronym: OmegaMI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Only 5 individuals were able to be recruited.
Sponsor: University of Rochester (Other)
Collaborators: GlaxoSmithKline (Industry); Albany College of Pharmacy and Health Sciences (Other)
Responsible Party: Principal Investigator, Robert Block, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVZ114193
Record Dates: First submitted 2010-06-25; First posted 2010-07-01 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Infarction
Keywords: Acute Coronary Syndrome; Fish Oils; Platelet Function Tests; Cardiac Electrophysiology
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome | interventions — Omacor; Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovaza® (Experimental): Lovaza® is a prescription grade EPA+DHA fish oil supplement. Four capsules (each containing 1 gram of fish oil) were taken within hours after the PCI, daily for the duration of hospitalization, and daily for 1 week until a post-discharge follow-up appointment.
  Interventions: Drug: Lovaza®
- Corn Oil (Placebo Comparator): The placebo contained 1 gram of corn oil in each capsule. Four capsules were taken within hours after the PCI, daily for the duration of hospitalization, and daily for 1 week until a post-discharge follow-up appointment.
  Interventions: Drug: The placebo contained 1 gram of corn oil in each capsule.

INTERVENTIONS:
Drug: Lovaza® — Lovaza® is prescription grade EPA+DHA fish oil supplement.
  Other Names: Fish oil
  Arms: Lovaza®
Drug: The placebo contained 1 gram of corn oil in each capsule. — Placebo Pill
  Other Names: Corn oil
  Arms: Corn Oil

SUMMARY:
This study will explore the safety and effectiveness of adding Lovaza® to the therapeutic program utilized internationally for the treatment of individuals with acute coronary syndromes.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease is the cause for over 19 million deaths in the US annually with coronary artery disease accounting for most of this mortality burden.1 Despite major advances in the treatment of coronary heart disease patients, a large number of victims of the disease who are apparently healthy die suddenly without prior symptoms. For those who arrive alive at an emergency department, a benefit is accrued from an orchestrated program of live-saving therapeutics designed to preserve ischemic or infarcted myocardium and prevent ventricular arrhythmias. However, despite improvements in door-to-balloon (angioplasty) times in the past decade, reductions in in-hospital mortality have not materialized.2 Average 30-day mortality from ST elevation MI has been shown to be approximately 7% despite the modern aggressive approach of utilizing acute pharmacologic and percutaneous interventions as well as a comprehensive approach to risk factor modification.3 Antiplatelet agents including aspirin, clopidogrel, heparin, and IIb/IIIa inhibitors represent stalwart components of the acute coronary syndrome therapeutic treatment program. At the same time, the safety of combination antiplatelet agents used acutely and chronically in individuals with an acute coronary syndrome is concerning as bleeding complications can result in serious, life-threatening consequences.4 Studies have shown that patients treated with the combination of aspirin and clopidogrel have a small but significant increased risk of major and minor bleeding compared to each agent alone.4-6 In contrast, the use of fish oil in conjunction with aspirin and clopidogrel in patients with cardiovascular disease followed for an average of 33 months has been shown to have no significant effect on risk of major and minor bleeding compared to those on aspirin and clopidogrel alone, with a trend toward a reduced risk of minor bleeding in those taking fish oil.4 In Preliminary Data it is shown that a robust synergistic effect between Lovaza® and aspirin on the downregulation of platelet function may occur. These data suggest that the most potent omega-3 fatty acids found in fish oil (eicosapentaenoic acid {EPA} and docosahexaenoic acid {DHA}) act acutely to modulate a major contributor to the pathophysiology of acute coronary syndromes. This study will randomize 60 patients with ST elevation myocardial infarction to treatment with Lovaza® or placebo and measure the differences in platelet function and electrophysiologic parameters between treatment arms during their acute hospitalization and 1 week after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction documented by at least 2 of the following:

  1. Typical symptoms
  2. Abnormal levels of cardiac biomarkers (troponin I or T or CK-MB mass) with at least one determination > 99th percentile or ULN for the laboratory
  3. ECG findings diagnostic of myocardial infarction based on the American College of Cardiology criteria.
* Status-post urgent or emergent PCI
* Have a Thrombolysis In Myocardial Infarction (TIMI) flow grade = 3 (complete perfusion) post PCI.
* Have the capacity for informed consent (e.g. without significant dementia or sedation from medication)
* Ingested 325 mg of chewed aspirin as part of the acute coronary syndrome treatment protocol.

Exclusion Criteria:

* No informed consent
* Daily aspirin use prior to index hospitalization
* Known prior myocardial infarction
* Known pregnancy
* Known allergy to fish, fish oil, or aspirin
* Known active internal or non-superficial bleeding, known bleeding disorder, coagulation defect, or thrombocytopenia
* Thrombolysis in the past 12 hours
* Treatment with a IIbIIIa inhibitor during index hospitalization
* Cardiogenic shock or symptomatic hypotension or sitting SBP < 95 mmHg
* Severe uncontrolled hypertension (≥180/110) or hypertensive retinopathy
* A history of major surgery, trauma, retinal hemorrhage, significant gastrointestinal (not hemorrhoidal) or genitourinary bleeding in the past 6 weeks
* A history of cerebrovascular attack within two years, or cerebrovascular attack with a significant residual neurological deficit
* A known arteriovenous malformation or aneurysm
* Severe liver insufficiency (ALT ≥ 3 times normal)
* Renal insufficiency requiring dialysis
* A known diagnosis of vasculitis
* Participation in another clinical study
* History of malignancy, except subjects who have been disease-free for greater than 10 years, or whose only malignancy has been basal or squamous cell skin carcinoma
* Oral contraceptive use
* Daily use of NSAIDs
* History of drug or alcohol abuse, or current weekly alcohol consumption >14 units/week (1 unit = 1 beer, 1 glass of wine, 1 mixed cocktail containing 1 shot of alcohol)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Block, MD, MPH, Principal Investigator — University or Rochester
Locations (1):
- University or Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Corn Oil: The placebo contained 1 gram of corn oil in each capsule. Four capsules were taken within hours after the PCI, daily for the duration of hospitalization, and daily for 1 week until a post-discharge follow-up appointment.
  The placebo contained 1 gram of corn oil in each capsule. : Placebo Pill
- Lovaza®: Lovaza® is a prescription grade EPA+DHA fish oil supplement. Four capsules (each containing 1 gram of fish oil) were taken within hours after the PCI, daily for the duration of hospitalization, and daily for 1 week until a post-discharge follow-up appointment.
  Lovaza® : Lovaza® is prescription grade EPA+DHA fish oil supplement.
Period: Overall Study
Arm/Group | Corn Oil | Lovaza®
Started | 0 (We did not complete the study.) | 4 (We did not complete the study.)
Completed | 0 (We did not complete the study.) | 4 (We did not complete the study.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corn Oil | Lovaza® | Total
Number analyzed (Participants) | 0 | 4 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 3 | 3
  >=65 years |  | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 60.25 (10) | 60.25 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Platelet Function
Description: Platelet function will be measured with PFA-100 test which has been shown to correlate with an increased risk for cardiovascular events in several well conducted studies and in a meta-analysis. The PFA-100 measures the number of seconds required for a clot to form in whole blood which is passed through an aperture in a cartridge coated with epinephrine. It is meant to imitate clotting in human arteries.
Time Frame: 12 hours
Population: We did not complete the study and no subjects were randomized to corn oil
Measure: Mean (Full Range); unit: seconds
Arm/Group | Corn Oil | Lovaza®
Number analyzed (Participants) | 0 | 4
seconds |  | 130.25 [101 to 190]

2. Secondary Outcome: Cardiac Electrophysiology
Description: A 20-minute supine 12-lead Holter ECG will allow the quantification of a series of standard ECG parameters as well as provide insight into frequency-domain HRV parameters, QRS duration and morphology, using signal-averaged ECG (SAECG), repolarization morphology, and variability utilizing specialized programs.
Time Frame: 1 week
Population: Data was not collected for this outcome measure.
Arm/Group | Corn Oil | Lovaza®
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Corn Oil | Lovaza®
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4

LIMITATIONS AND CAVEATS:
no adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No